CLINICAL TRIAL: NCT02163785
Title: Estudio A.P.PRO: Estrategia quirúrgica en la amputación Abdominoperineal cilíndrica Del Recto Por cáncer: posición de litotomía vs. Prono-navaja
Brief Title: Abdominoperineal Extra-Elevators Rectal Resection for Cancer: Prone Position vs. Supine Position
Acronym: APPRO
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: insufficient recruitment rate
Sponsor: Hospital Universitario La Fe (Other)
Collaborators: Fundacion Para La Investigacion Hospital La Fe (Other); Instituto de Salud Carlos III (Other Government)
Responsible Party: Principal Investigator, Matteo Frasson, MD, PhD, Hospital Universitario La Fe
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: APPRO
Record Dates: First submitted 2014-06-12; First posted 2014-06-16 (Estimated); Last update posted 2021-10-01 (Actual); Status verified 2021-09

CONDITIONS: Rectal Cancer; Abdominoperineal Resection
Keywords: Inferior rectal cancer; Abdominoperineal resection; Miles operation; Supine Miles operation; Prone Miles operation; Total mesorectal excision; Circumferential radial margin
MeSH Terms: conditions — Rectal Neoplasms | interventions — Proctectomy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Supine position (Active Comparator): Abdominoperineal resection - perineal time- in supine position
  Interventions: Procedure: Abdominoperineal extra-elevators rectal resection for low lying rectal cancer
- Prone position (Experimental): Abdominoperineal resection - perineal time- in prone position
  Interventions: Procedure: Abdominoperineal extra-elevators rectal resection for low lying rectal cancer

INTERVENTIONS:
Procedure: Abdominoperineal extra-elevators rectal resection for low lying rectal cancer — Abdominoperineal extra-elevators rectal resection for low lying rectal cancer involving anal sphincter complex
  Other Names: Abdominoperineal resection of the rectum; Abdominoperineal excision of the rectum; Abdominoperineal resection

SUMMARY:
Prospective multicenter randomized controlled trial comparing the prone vs. the supine position of the perineal time of the Miles operation in patients with advanced rectal cancer.

Primary objective:

- Pathological circumferential resection margin

Secondary objectives:

* 5 year oncological outcomes
* Morbimortality rates
* Surgical specimen quality
* Perineal hernia incidence

ELIGIBILITY:
Inclusion Criteria:

* Patients with primary low lying rectal cancer involving or threatening anal sphincter complex as seen in MRI

Exclusion Criteria:

* American Society of Anaesthesiologists classification of Physical Health (ASA) IV patients
* Locally palliative purpose of the operation
* Age < 18 years
* Preoperative indication for pelvic exenteration
* Pregnancy
* Lack of patients consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2014-06; Primary Completion 2021-01 (Actual); Study Completion 2021-01 (Actual)

PRIMARY OUTCOMES:
Assessment of the circumferential resection margin | 15-30 days after surgery date
  Histopathological report of the circumferential resection margin of the surgical specimen obtained in patients that underwent perineal time of Miles procedure in prone vs supine position.

SECONDARY OUTCOMES:
Histopathological quality of surgical specimen | 15-30 days after
  Comparison of the quality of the surgical specimen in terms of integrity of the circumferential resection margin, accidental iatrogenic rupture etc.

OTHER OUTCOMES:
Oncological outcomes | 5 years
  Compare the incidence of local oncological disease, distance metastasis and survival in a 5 year follow up time span.
Morbidity of the perineal incision. | 1 day, 60 days ,1 ,2,3,4 and 5 years after surgery
  Evaluation the clinical outcome of the perineal wound in terms of infection, dehiscence, perineal hernia etc.

CONTACTS AND LOCATIONS:
Overall Officials: Matteo Frasson, MD, PhD, Principal Investigator — Hospital Universitario y Politecnico La Fe; Eduardo Garcia-Granero, MD, PhD, EBSQ-c, Study Chair — Hospital Universitario y Politecnico La Fe
Locations (19):
- Spain (19):
  - Hospital Universitario Reina Sofia, Córdoba, Andalusia
  - Hospital del SAS, Jerez de la Frontera, Andalusia
  - Hospital Universitario Donostia, Donostia / San Sebastian, Basque Country
  - Hospital General, Medina del Campo, Castille and León
  - Hospital Bellvitge, Barcelona, Catalonia
  - Hospital del Mar, Barcelona, Catalonia
  - Hospital Universitario Josep Trueta, Girona, Catalonia
  - Hospital Universitario Parc Tauli, Sabadell, Catalonia
  - Complexo Hospitalario Universitario, Ourense, Galicia
  - Complejo Hospitalario Universitario, Vigo, Galicia
  - Complejo Hospitalario, Pamplona, Navarre
  - Hospital General Universitario, Elche, Valencia
  - Hospital General, Requena, Valencia
  - Hospital de Sagunto, Sagunto, Valencia
  - Hospital Luis Alcanyis, Xàtiva, Valencia
  - Hospital Universitario "Virgen de la Arrixaca", Murcia
  - Hospital Universitario y Politecnico La Fe, Valencia
  - Hospital Arnau de Vilanova, Valencia
  - Hospital Clinico Universitario, Valencia

REFERENCES:
- [Background] Garcia-Granero E, Faiz O, Munoz E, Flor B, Navarro S, Faus C, Garcia-Botello SA, Lledo S, Cervantes A. Macroscopic assessment of mesorectal excision in rectal cancer: a useful tool for improving quality control in a multidisciplinary team. Cancer. 2009 Aug 1;115(15):3400-11. doi: 10.1002/cncr.24387. PMID 19479978
- [Background] Heald RJ, Moran BJ, Ryall RD, Sexton R, MacFarlane JK. Rectal cancer: the Basingstoke experience of total mesorectal excision, 1978-1997. Arch Surg. 1998 Aug;133(8):894-9. doi: 10.1001/archsurg.133.8.894. PMID 9711965
- [Background] Flor-Lorente B, Frasson M, Montilla E. Extralevator abdominoperineal resection in the prone position. Cir Esp. 2014 Mar;92 Suppl 1:30-9. doi: 10.1016/S0009-739X(14)70006-5. English, Spanish. PMID 24842689
- [Derived] Frasson M, Garcia-Granero E. Reply to Kelly et al. Colorectal Dis. 2016 Mar;18(3):312-3. doi: 10.1111/codi.13272. No abstract available. PMID 26757199